CLINICAL TRIAL: NCT01010152
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Comparative Bioavailability Study fo Codeine 30 mg Tablets and Tylenol #3 Tablets Under Fasting Conditions
Brief Title: Comparative Bioavailability Study of Codeine Sulfate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CODE-T30-PVFS-1
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O(6)-codeine methyl ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Codeine Sulfate (Experimental): 30 mg tablet
  Interventions: Drug: Codeine Sulfate
- Tylenol #3 (Active Comparator): 30 mg tablet
  Interventions: Drug: Codeine Sulfate

INTERVENTIONS:
Drug: Codeine Sulfate — 30 mg Tablet
  Other Names: Tylenol #3 Tablets

SUMMARY:
The objective of this study was to assess the comparative bioavailability of codeine from Roxane Laboratories' Codeine Sulfate 30mg tablets to Tylenol® #3 (acetaminophen 300mg with codeine phosphate 30mg) under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to codeine sulfate or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick Bieberdorf, M.D., Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research LLC, San Antonio, Texas, United States